CLINICAL TRIAL: NCT03063983
Title: A Study Multicenter Randomized to Assess the Efficacy and Toxicity of Adding Metronomic Therapy to the Standard Treatment of Patients With High Grade Malignant Osteosarcoma With Metastatic Lung Disease at Diagnosis and Primary Resectable Tumor: A Study by the Latin American Group for Treatment of Osteosarcoma
Brief Title: Clinical Trial Evaluating Metronomic Chemotherapy in Patients With Metastatic Osteosarcoma
Acronym: GLATO2017
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Apoio ao Adolescente e a Crianca com Cancer (Other)
Responsible Party: Principal Investigator, Antônio Sérgio Petrilli, Principal Investigator, Grupo de Apoio ao Adolescente e a Crianca com Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLATO2017
Record Dates: First submitted 2017-01-27; First posted 2017-02-24 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; metastatic; metronomic therapy
MeSH Terms: conditions — Osteosarcoma; Neoplasm Metastasis | interventions — Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maintenance therapy (Experimental): 104 weeks of continuous oral low dose chemotherapy with cyclophosphamide (CPM) and methotrexate (MTX) following 31 weeks of MAP
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate
- Control (No Intervention): 31 weeks of MAP

INTERVENTIONS:
Drug: Cyclophosphamide — Continuous oral cyclophosphamide
  Arms: Maintenance therapy
Drug: Methotrexate — Continuous oral methotrexate
  Arms: Maintenance therapy

SUMMARY:
Preclinical models show that a daily antiangiogenic regimen at low-dose may be effective against chemotherapy-resistant tumors. The aim of this study is to evaluate the efficacy of maintenance therapy with continuous oral cyclophosphamide and methotrexate in patients with high grade, operable, metastatic osteosarcoma (OST) of the extremities. The primary end point is event-free survival (EFS) from randomization

DETAILED DESCRIPTION:
The study design includes backbone of 10 weeks of preoperative therapy using MAP (high-dose methotrexate, cisplatin, doxorubicin and dexrazoxane). Metastatic patients were randomized to high-dose chemotherapy for 31 weeks (arm 1) or concomitant metronomic therapy (MTX plus cyclophosphamide) such as 31 weeks of high-dose chemotherapy, followed by 73 weeks of metronomic therapy after completion of high-dose chemotherapy, totaling 104 weeks of metronomic therapy (arm 2).

ELIGIBILITY:
Inclusion Criteria:

* A newly diagnosed patient, previously untreated, with a high degree of malignancy, confirmed by biopsy. Participant with OST as a neoplasm are also eligible
* Participant with staging imaging studies performed less than four weeks. Otherwise, it should be re-staged
* If pre-chemotherapy amputation is necessary, the participant will enter the study being excluded from the evaluation of tumor necrosis grade according to Huvos, but eligible for survival analysis
* Participant aged ≥ 16 years should have a Karnofsky performance score> 50 or WHO / ECOG ≥ 2 and patients <16 years should have a Lansky performance score> 50. Participant with a performance score impaired by the presence of a pathological fracture are eligible
* Patients with normal organic function
* Sexually active participant should agree to use contraceptive methods throughout the treatment
* Female participant should have a negative pregnancy test

Exclusion Criteria:

* If the participant or their legal guardian refuses to sign the informed consent form / consent term it will not be included in the study.

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-01-02 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and toxicity of adding metronomic therapy in disease event-free survival. | Five years
  To assess the impact of adding metronome therapy to the standard treatment of patients with resectable end-stage osteosarcoma and metastatic lung disease in event-free survival.

SECONDARY OUTCOMES:
Efficacy and toxicity of adding metronomic therapy in overall survival | Five years
  To evaluate the impact of the addition of metronomic therapy to the standard treatment of patients with end-resectable osteosarcoma and metastatic lung disease in overall survival.
Cardiotoxicity (occurrence of cardiotoxicity) | Five years
  To compare the occurrence of cardiotoxicity with the addition of dexrazoxane since the first cycle of doxorubicin with the findings of the previous study (GLATO 2006).
Immunohistochemistry (expression of VEGF) | Five years
  Immunohistochemistry the expression of VEGF in the biopsy, primary tumor and metastases

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia F Fontes, Study Chair — Grupo de Apoio ao Adolescente e a Crianca com Cancer
Locations (1):
- Grupo de Apoio ao Adolescente e a Criança com Câncer, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided